CLINICAL TRIAL: NCT06659991
Title: JIT: Effects of Pain on Laboratory Drinking Topography and Daily Drinking in People With Chronic Temporomandibular Disorder (TMD) Pain
Brief Title: JIT: Effect of Pain on DT in TMD
Acronym: TMD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ANES-2024-33184
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Temporomandibular Disorder (TMD)
Keywords: alcohol; temporomandibular disorder (TMD); chronic pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Chronic Pain | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: This is a crossover design wherein participants consume either alcohol-containing beverages (beer or cider) or sparkling water over two laboratory sessions.
Masking Description: This study does not employ masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- TMD Group 1 (Experimental): People with an established diagnosis of temporomandibular disorder (TMD) assigned to Ethanol intervention
  Interventions: Drug: alcohol condition
- TMD Group 2 (Sham Comparator): People with an established diagnosis of temporomandibular disorder (TMD) assigned to sparkling water (control)
  Interventions: Other: control condition
- Pain-free Control Group 1 (Experimental): People without an established diagnosis of temporomandibular disorder (TMD) or other chronic pain condition assigned to Ethanol intervention
  Interventions: Drug: alcohol condition
- Pain-free Control Group 2 (Sham Comparator): People without an established diagnosis of temporomandibular disorder (TMD) or other chronic pain condition assigned to sparkling water (control)
  Interventions: Other: control condition

INTERVENTIONS:
Drug: alcohol condition — Ethanol
  Arms: Pain-free Control Group 1; TMD Group 1
Other: control condition — sparkling water
  Arms: Pain-free Control Group 2; TMD Group 2

SUMMARY:
Individuals with chronic temporomandibular disorder (TMD) pain are at increased risk for alcohol-related consequences compared to those without pain, and growing evidence suggests pain is a potent motivator for alcohol use in many individuals. However, few systematic examinations of modifiable and non-modifiable risk factors, including orofacial pain status, have been conducted. This project addresses this gap in knowledge by determining the effect of pain on drinking topography in heavy drinkers with and without chronic TMD pain in both the laboratory and daily life.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study must be 21 years to 65 years of age and provide a driver's license or other state-issued ID.
* Participants must also be sufficiently fluent in English to provide informed consent and understand questionnaires and instructions for laboratory procedures.
* Participants must report drinking of, on average, at least 1 drink 3 days/week over the past 6 months.
* Meet Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for myalgia (masticatory muscle pain), arthralgia (TMJ pain), or a combination (Schiffman et al., 2014) (TMD group only).
* Own a smartphone with internet access.
* Use of prescription medications will be allowed, provided they do not contraindicate alcohol use.

Exclusion Criteria:

* Use of opioid analgesics within the past month;
* Current major depression;
* History of any psychotic disorder;
* Under-controlled hypertension or diabetes (as reflected by self-report); neurological disease (e.g., multiple sclerosis, epilepsy, amyotrophic lateral sclerosis, Parkinson's disease);
* Serious medical illness (e.g., hepatitis, HIV/AIDS);
* Impaired cognitive function;
* History of substance use disorder (including nicotine/tobacco);
* Alcohol naïve
* Alcohol use disorder, or currently attempting to quit or cut down on using alcohol
* Positive pregnancy test
* Breastfeeding or intending to become pregnant
* Loss of sensation in the lower leg
* Inability to complete study tasks due to weakness, immobilization, or loss of limbs
* Chronic pain (Control group only)
* A urine-based drug screen for tetrahydrocannabinol, cocaine, benzodiazepines, morphine, and methamphetamine (Innovacon, Inc., San Diego, CA) will be performed. Participants testing positive for any substance will be discontinued.
* Medications that contraindicate alcohol use

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2029-09-07 (Estimated); Study Completion 2029-09-07 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use Topography | 30 minutes
  Variables reflecting microstructure of alcohol use during self-administration, including sip interval and sip volume.
Heat Pain Intensity | 30 minutes
  Pain intensity of heat stimuli applied during self- administration sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Boissoneault, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States